CLINICAL TRIAL: NCT04243902
Title: Urinary Catheter 'Fill and Flush' Valve: Safety, Effectiveness, Acceptability and Feasibility Trial
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: No participants met all the inclusion criteria required within the recruitment time period
Sponsor: University of Southampton (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); BlueWind Medical (Industry); University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Device Feasibility
Other Study IDs: 41448; 245818 (Other: IRAS)
Record Dates: First submitted 2019-08-21; First posted 2020-01-28 (Actual); Last update posted 2023-10-06 (Actual); Status verified 2023-10

CONDITIONS: Indwelling Urinary Catheter Users
Keywords: urinary catheter; IDC

STUDY DESIGN:
Intervention Model Description: 2 groups, 1 group including interim safety review
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1 - standard manual valve (without leg-bag) (Experimental): The valve will initially be tested in 8 participants who currently use a standard manual valve (without leg-bag).
  This first group will include a safety cohort of participants (n=4). All safety data will be reviewed from the initial 4 participants before further participants can undergo the study investigation.
  Interventions: Device: Fill and Flush Valve
- 2 - drainage bag with free drainage (Experimental): The valve will then be tested with participants (n=8) who currently use a drainage bag with free drainage.
  Interventions: Device: Fill and Flush Valve

INTERVENTIONS:
Device: Fill and Flush Valve — The fill and flush valve (Figure 1) is an automated valve which is designed to open in response to rising bladder pressure which occurs as the bladder becomes full. The valve is situated between the IDC and the drainage bag as a manual valve would be.
  There are three variants of the valve which respond to different degrees of bladder pressure. People's bladders function at different pressure levels. One of the aims of this study is to gain preliminary data on which valve variant works and under which circumstances. Pressure ranges are as follows:
  Low: 22 - 49cm H2O Medium: 35 - 61cm H2O High: 53 - 79cm H2O
  Other Names: EM02, EM03, EM04

SUMMARY:
The fill and flush valve (valve) is an automated valve which is designed to open in response to rising bladder pressure which occurs as the bladder becomes full. The valve is situated between the IDC and the drainage bag as a manual valve would be.

DETAILED DESCRIPTION:
The objective of this study is to assess preliminary safety, effectiveness, reliability, comfort and user acceptability of the valve with adults who have a long-term IDC and the feasibility of undertaking future community-based evaluation.

To do this the investigators will

* determine if the valve functions reliably i.e. automatically opens to drain urine within acceptable individual bladder volumes with a range of patients;
* determine if the valve functions effectively i.e. allows for the complete bladder emptying (< 100ml post void residual) during rest and daily activities;
* determine if the process of filling and automatic draining is comfortable and acceptable for participants;
* collect preliminary data on the potential for bioburden/biofilm following in human use of the valve;
* assess the feasibility of undertaking a future randomised control trial of the valve.

Group 1 - The investigators will test the valve with participants (n=8) who currently use a standard manual valve (without leg-bag).This first group will include a safety cohort of participants (n=4). All safety data will be reviewed from the initial 4 participants before further participants can undergo the study investigation.

Group 2- The Investigators will test the valve with participants (n=8) who currently use a drainage bag with free drainage.

The data collection process and study procedures will be identical for both groups.

After use(in both groups), the valves will be examined microbiologically in the University of Southampton laboratory to detect bioburden and/or biofilm to ascertain a baseline for future studies.

ELIGIBILITY:
Inclusion Criteria:

* IDC-users (urethral or suprapubic), over 18, who have had a catheter in situ for at least one month and use a manual valve or drainage bag to collect urine
* Independent with catheter care needs (e.g. bag emptying or valve opening)
* Able to transfer from bed to chair, stand and walk short distances unaided
* Able to drink moderate levels of fluid (500mls in the first 2 hours and 150mls per hour thereafter)
* Able to provide informed consent (self-report and research nurse assessment)
* Usual medical provider provides confirmation of suitability

Exclusion Criteria:

* End stages of a terminal illness
* Current treatment of urinary tract infection
* Has been advised by a urologist against using a valve on clinical grounds
* Lack of bladder sensation (e.g. unable to sense when bladder needs emptying)
* Previous bladder surgery that could affect the integrity of the bladder
* At known risk of autonomic dysreflexia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-02-13 (Actual); Primary Completion 2023-07-18 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
Safety: Reliability | An average of 16 hours in total
  Valve opening - Proportion of observations of automatic valve opening before bladder capacity (500ml or less) is reached - as measured by bladder scanner
Safety: Effectiveness | An average of 16 hours in total
  Bladder emptying - proportion of valve voids with residual urine <100ml - as measured by bladder scanner.
Safety: Effectiveness | An average of 16 hours in total
  Bladder emptying - Participant report (Valve self-report questionnaire)
Comfort | An average of 16 hours in total
  Participant report (Valve self-report questionnaire)

SECONDARY OUTCOMES:
User acceptability | An average of 16 hours in total
  Valve self-report questionnaire (Valve self-report questionnaire)
User acceptability | An average of 16 hours in total
  EQ-5D-5L
User acceptability | An average of 16 hours in total
  Long-term Catheter Quality of Life Tool

CONTACTS AND LOCATIONS:
Overall Officials: Cathy Murphy, Principal Investigator — University of Southampton
Locations (1):
- University Hospital Southampton, Southampton, Hampshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No